CLINICAL TRIAL: NCT04830020
Title: Use of Inhaled High-molecular Weight Hyaluronan in Patients With Severe COVID19: Feasibility and Outcomes
Acronym: HA-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CampusBioMedico; 1ZIDES102465 (NIH)
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMW-HA (Active Comparator): HMW-HA (Yabro - 5 ml of saline containing 0.3% hyaluronic acid sodium salt)
  Interventions: Drug: HMW-HA
- placebo (Placebo Comparator): 5 ml of saline via nebulizer b.i.d.
  Interventions: Drug: HMW-HA

INTERVENTIONS:
Drug: HMW-HA — Aerolized administration b.i.d.
  Other Names: Yabro

SUMMARY:
To determine whether inhaled Yabro protects against progression of COVID19-induced respiratory failure preventing the passage to non-invasive ventilation (NIV) and promotes recovery from COVID19 lung disease in hospitalized patients.

DETAILED DESCRIPTION:
All patients will be treated with state of the art COVID19 treatment as per the treating clinician (Remdesivir, systemic corticosteroids, monoclonal antibodies, convalescent plasma, biologic cytokine inhibitors and other interventions as per the latest guidelines). Patients randomized to the active intervention group will also receive HMW-HA (Yabro®, 5 ml of saline containing 0.3% hyaluronic acid sodium salt) via nebulizer, while patients randomized in the control group will receive a matching placebo two times daily.

Due to increased risk for SARS-CoV-2 transmission via the usual mask nebulization procedure, patients will receive the nebulized treatment via high-flow oxygen tubing as described in the literature 36-38. Patients will be treated until there is a qualitative change in oxygen requirement, i.e. either progression to assisted ventilation (non-invasive or invasive), or weaning from oxygen supplementation. Because COVID19 may result in long-term O2 dependency, the study and treatment period will be limited to a maximum of 10 days.

Moreover, a blood sample (20 ml) will be taken at baseline and after 10 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Diagnosis of COVID19 by validated SARS-CoV-2 antigen, RT-PCR, or other molecular diagnostic assay, using an appropriate sample such as NP, nasal, oropharyngeal [OP], or saliva) and no alternative explanation for current clinical condition.
* Respiratory failure requiring oxygen therapy
* Has symptoms consistent with COVID-19, and is in non-fibroproliferative stage of disease, as determined by investigator.

Exclusion Criteria:

* Respiratory arrest or the need for immediate intubation;
* Upper airway obstruction;
* Facial trauma;
* Inability to cooperate (e.g. agitation or dementia)
* Inability to give informed consent
* Participation in another study for COVID19 treatments
* Deterioration due to other reasons than progressive COVID19 pneumonia per clinical judgment, e.g. pulmonary thromboembolism, heart failure, renal failure etc.
* Palliative care or expectation that patient will not survive > 72 hours post randomization per clinical judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Cumulative time on oxygen | 10 days
  cumulative duration of oxygen treatment

SECONDARY OUTCOMES:
Need for advanced airway intervention or death due to COVID19; | 10 days
  need of intubation or death due to COVID19
Rate of change of respiratory rate; | 10 days
  rapidity of decrease of respiratory rate
Change in PaO2 /FiO2 ratio during treatment | 10 days
  improvement of PaO2/FiO2 ratio after 10 days of treatment
Time to discharge from hospital | 10 days
  decrease of cumulative days of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Antonelli Incalzi, MD, Principal Investigator — Università Campus-Biomedico di Roma
Locations (1):
- Università Campus Biomedico di Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No